CLINICAL TRIAL: NCT00812422
Title: Multi-center, Randomized, Double Blinded (Double-dummy), Active-Controlled Parallel-group Comparative, Phase 3 Clinical Trial to Assess the Efficacy and Safety of Dexibuprofen Syrup Compared to Ibuprofen Syrup in Patients With Fever of Common Cold (Acute Upper Respiratory Infection)
Brief Title: The Efficacy and Safety of Dexibuprofen Syrup
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Inje University (Other)
Responsible Party: Chang-Keun Kim, Inje University Sanggye Paik Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AG_DIBU_2007
Record Dates: First submitted 2008-12-19; First posted 2008-12-22 (Estimated); Last update posted 2010-01-18 (Estimated); Status verified 2010-01

CONDITIONS: Fever; Respiratory Tract Infection
Keywords: Fever due to acute upper respiratory tract infection
MeSH Terms: conditions — Fever; Respiratory Tract Infections | interventions — dexibuprofen; Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Dexibuprofen 1 (Experimental): Dexibuprofen 2.5 or 5 mg/kg
  Interventions: Drug: Dexibuprofen
- Dexibuprofen 2 (Experimental): Dexibuprofen 3.5 or 7 mg/kg
  Interventions: Drug: Dexibuprofen
- Ibuprofen (Active Comparator): Ibuprofen 5 or 10 mg/kg
  Interventions: Drug: Ibuprofen

INTERVENTIONS:
Drug: Dexibuprofen — one dose of Dexibuprofen 2.5 or 5 mg/kg
  Arms: Dexibuprofen 1
Drug: Dexibuprofen — one dose of Dexibuprofen 3.5 or 7 mg/kg
  Arms: Dexibuprofen 2
Drug: Ibuprofen — one dose of Ibuprofen 5 or 10 mg/kg
  Arms: Ibuprofen

SUMMARY:
The purpose of this study is to compare the safety and efficacy of dexibuprofen syrup and ibuprofen syrup in patients with fever due to common cold.

ELIGIBILITY:
Inclusion Criteria:

* Common cold with fever
* Age 6 months to 14 years

Exclusion Criteria:

* Gastric ulcer
* Bleeding tendency
* Liver disease
* Kidney disease
* Hypertension
* Hypersensitivity to the drug

Ages: 6 Months to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 260 (Actual)
Dates: Start 2008-02; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
measure reduction in fever | measure temperature every hour for 3 hours then once again 3 days later

SECONDARY OUTCOMES:
determine safety of dexibuprofen by unwanted reaction, clinical laboratory test and physical examination. | every hour for 3 hours (unwanted reaction). 3 days later (clinical laboratory test and physical examination).

CONTACTS AND LOCATIONS:
Overall Officials: Young Yull Koh, Study Director — Seoul National University Hospital; Chang-Keun Kim, Principal Investigator — Inje University
Locations (4):
- South Korea (4):
  - Asan Medical Center, Seoul
  - Inje University Sanggye Paik Hospital, Seoul
  - Korea University Hospital, Seoul
  - Kyung Hee University Hospital, Seoul